CLINICAL TRIAL: NCT02241577
Title: Surgical and Non-surgical Treatment of Peri-implantitis: Multi-center Randomised Controlled Trial of 12-months Follow-up
Brief Title: Surgical and Non-surgical Treatment of Peri-implantitis
Acronym: Perio-implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGSimplant2014; CNPq14_2013 (Other Grant/Funding Number: CNPq (Brazilian Counsel for Research))
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Peri-implantitis
Keywords: peri-implantitis; dental implants; randomized controlled trial; non-surgical periodontal treatment; will be defined by the presence of alveolar bone loss of at least 3mm, pocket depth of at least 5mm and bleeding on probing.
MeSH Terms: conditions — Peri-Implantitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Experimental): Surgical access for scaling and disinfection of dental implant
  Interventions: Procedure: Surgical treatment
- Non-surgical treatment (Experimental): Non-surgical subgingival scaling and disinfection of dental implant
  Interventions: Procedure: Non-surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Flap surgery around dental implant for scaling and disinfection of the titanium surface under local anesthesia
  Arms: Surgical treatment
Procedure: Non-surgical treatment — Non-surgical subgingival scaling and disinfection of the titanium surface of dental implant under local anesthesia
  Arms: Non-surgical treatment

SUMMARY:
This study will compare surgical and non surgical treatments of peri-implantitis. Peri-implantitis is an inflammation around dental implants that can lead to the loss of the implant over time if no treatment is established. The signs of peri-implantitis included bleeding of the gingiva, swelling and redness. Most of times there is no pain. Patients presenting with these characteristics will be included at random to one of the treatment groups. Those allocated to the non-surgical group will received implant cleansing after local anesthesia using adequate instruments. In the surgical group, patients will be submitted to a surgical procedure around the implant for visualization and cleansing also after local anesthesia. All patients will be followed over a 12-month period. The hypothesis is that surgical treatment is better than non-surgical treatment regarding clinical, radiographic, microbiological, and immunological.characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with at least one dental implant with peri-implantitits
* Individuals with good general health conditions;
* Individuals presenting at least 10 natural teeth;
* Individuals with no signs of active periodontitis

Exclusion Criteria:

* Individuals who received periodontal treatment in the last three months
* Pregnant
* Systemic condition that interferes with treatment such as diabetes
* Individuals who are taking or have taken antibiotics or anti-inflammatory medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Pocket depth reduction | 12 months

SECONDARY OUTCOMES:
Clinical attachment level changes | 12 months
Alveolar bone level changes | 12 months
Subgingival microbiota changes | 12 months
Gingival crevicular fluid immune-inflammatory biomarkers | 12 motnhs
Serum biomarkers of inflammation | 12 months
Bleeding on probing | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano K Rosing, PhD, Study Chair — Federal University of Rio Grande do Sul; Joao Augusto P Oliveira, MS, Principal Investigator — Federal University of Rio Grande do Sul; Tassiane P Wagner, DDS, Principal Investigator — Federal University of Rio Grande do Sul; Fernando S Rios, MS, Principal Investigator — Federal University of Rio Grande do Sul; Ricardo SA Costa, MS, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Alex Haas, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Site of the School of Dentistry — http://www.ufrgs.br/odonto
- See also: Site of the Post-graduate Program in Dentistry — http://www.ufrgs.br/ppgodo/index.php